CLINICAL TRIAL: NCT06093594
Title: Understanding Patient Engagement Trends in Stage IV Melanoma Clinical Trials
Brief Title: Investigating Participation Patterns Among Stage IV Melanoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 74815433
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stage IV Melanoma
Keywords: Stage IV Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials, specifically focused on stage IV melanoma, are crucial in assessing the safety and efficacy of new treatments for this disease. These trials serve as fundamental instruments in determining whether emerging medications outperform standard therapies, providing compelling evidence to support wider implementation.

The main goal is to thoroughly scrutinize trial completion rates and voluntary withdrawals among this particular group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Diagnosis of stage IV melanoma
* Able to comprehend the investigational nature of the protocol and provide informed consent

Exclusion Criteria:

* Female patients who are currently pregnant or nursing
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IV melanoma who are actively considering enrolling in a clinical study for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of stage IV melanoma patients who decide to enroll in a clinical research | 3 months
Rate of stage IV melanoma patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scott JF, Conic RZ, Thompson CL, Gerstenblith MR, Bordeaux JS. Stage IV melanoma of unknown primary: A population-based study in the United States from 1973 to 2014. J Am Acad Dermatol. 2018 Aug;79(2):258-265.e4. doi: 10.1016/j.jaad.2018.03.021. Epub 2018 Mar 23. PMID 29580859
- [Background] Wevers KP, Hoekstra HJ. Stage IV melanoma: completely resectable patients are scarce. Ann Surg Oncol. 2013 Jul;20(7):2352-6. doi: 10.1245/s10434-013-2881-1. Epub 2013 Feb 8. PMID 23392854
- [Background] Luen S, Wong SW, Mar V, Kelly JW, McLean C, McArthur GA, Haydon A. Primary Tumor Thickness is a Prognostic Factor in Stage IV Melanoma: A Retrospective Study of Primary Tumor Characteristics. Am J Clin Oncol. 2018 Jan;41(1):90-94. doi: 10.1097/COC.0000000000000226. PMID 26325493

DOCUMENTS (1):
  • Informed Consent Form (2023-10-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT06093594/ICF_000.pdf